CLINICAL TRIAL: NCT02267642
Title: Efficacy and Safety of AbGn-168H in Patients With Active Psoriatic Arthritis: a 24-week, Open-label, Multi-center, Phase II Proof of Principle Trial.
Brief Title: A Phase II Study Evaluating the Efficacy and Safety of AbGn-168H in Patients With Active Psoriatic Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbGenomics B.V Taiwan Branch (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014.009.01
Record Dates: First submitted 2014-10-10; First posted 2014-10-17 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AbGn-168H (Experimental): Seven (7) intravenous doses of AbGn-168H on D1 (Week 0), Day 8 (Week 1), Day 15 (Week 2), Day D29 (Week 4), D43 (Week 6), Day 57 (Week 8) and Day 71 (Week 10)
  Interventions: Biological: AbGn-168H

INTERVENTIONS:
Biological: AbGn-168H — monoclonal antibody

SUMMARY:
To evaluate efficacy, safety, tolerability, and immunogenicity of AbGn-168H administered intravenously in patients with active psoriatic arthritis.

DETAILED DESCRIPTION:
This is an open-label, multi-center, multi-dose phase II proof of principle trial to study the efficacy and safety of AbGn-168H in patients with moderate to severe active psoriatic arthritis. A minimum of 15 patients and a maximum of 20 will be recruited in 1 dosing group. For safety evaluation, the parameters to be assessed include physical examination, vital signs (blood pressure, heart rate, respiratory rate and body temperature), 12-lead ECG, safety laboratory tests, adverse events and tolerability. For efficacy evaluation, patients will be evaluated for proportion of subject reaching American College of Rheumatology 20 (ACR 20) in week 12 and proportion of subjects reaching ACR 20, ACR 50 and ACR 70 at different time points; Disease Activity Score 28 (DAS28) at different time points, as well as Target Lesion Psoriasis Severity Score (TLPSS) and static Physician Global Assessment (sPGA) for subjects with active skin lesions at different time point.

ELIGIBILITY:
Inclusion criteria

1. Patient must give informed consent and sign an approved consent form prior to any study procedures
2. Age 18 to 75 (inclusive), males or females
3. Body weight < 140 kg
4. Subject has had a diagnosis of psoriatic arthritis for at least 6 months and currently meets the CASPAR criteria.
5. Patients must have moderate to severe active PsA at screening and baseline, defined as having greater than or equal to 3 tender (out of 68) and 3 swollen (out of 66) joints.
6. Patients must have at least one evaluable skin plaque, 2 cm in diameter, that can be followed with a target lesions score (scalp and groin lesions cannot be used), or documented psoriasis history.
7. Patients must have history of inadequate response or intolerance to NSAID or DMARD defined by the investigator.
8. If the patient is taking background corticosteroids, dose must be ≤ 10 mg/day prednisone (or equivalent) and must have been at a stable dose for at least 4 weeks prior to screening.
9. Use of nonsteroidal anti-inflammatory drugs (NSAIDs) for the treatment of psoriasis arthritis is permitted if the dose has been stable for at least 2 weeks prior to screening.
10. If the patient is taking methotrexate (MTX), the patient must have received methotrexate 7.5-25 mg/wk (p.o. or parenteral) for at least 12 weeks and at a stable dose for 4 weeks prior to screening. If the patient is not taking MTX, they must have been off the drug for at least 8 weeks prior to receiving the first dose (baseline).
11. Folic acid or folinic acid is required at least 1 mg per day or 5 mg per week for all patients taking MTX.
12. Whether or not the patient is taking methotrexate, all DMARDs (other than MTX) should be withdrawn at least 4 weeks prior to baseline (Visit 2) of first drug administration (4 weeks for etanercept, 8 weeks for infliximab, adalimumab, golimumab, certolizumab pegol and leflunomide, and 12 weeks for ustekinumab, c.f. Section 4.2.2). Subjects taking appremilast should discontinue the medication 2 weeks prior to receiving the first dose (baseline).
13. Females of childbearing potential must have a negative pregnancy test result prior to enrolment. Male and female of childbearing potential must agree to use a highly effective method of birth control during the study.

A female is considered of childbearing potential following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal ligation and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

A man is considered fertile after puberty unless permanently sterile by bilateral orchidectomy.

A highly effective method of birth control is defined as one which results in a low failure rate (less than 1% per year).

Exclusion criteria

1. History of malignancy in the past 5 years or suspicion of active malignant disease.
2. Evidence of current or previous clinically significant disease, medical condition other than psoriatic arthritis, or finding of the medical examination (including vital signs and ECG), that in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data. This criterion provides an opportunity for the investigator to exclude patients based on clinical judgment, even if other eligibility criteria are satisfied.
3. Presence of another rheumatic or skin disease that, in the opinion of the investigator, could confound the ability to discern response.
4. HIV infection or a known HIV-related Malignancy.
5. Chronic or acute hepatitis B and C, or carrier status.
6. History of recurrent significant infection; known active bacterial, viral, fungal, mycobacterial infection, or any major episode of infection requiring hospitalization or treatment with iv antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening.
7. Tuberculosis or a positive Quantiferon test for tuberculosis.
8. History of allergy/hypersensitivity to a systemically administered biologic agent or its excipients.
9. Intake of restricted medications (c.f. Section 4.2.2) or other drugs considered likely to interfere with the safe conduct of the study.
10. Previous treatment with any cell-depleting therapies, including investigational agents (e.g., CAMPATH, anti-CD4, anti-CD5, anti-CD3). Patients with Orencia or Toclizumab treatment within 8 weeks, IVIG, Natalizumab or Prosorba Column treatment within 6 months, and anti-CD19 or anti-CD20 treatment within 1 year should be excluded.
11. Immunization with a vaccine within 4 weeks prior to baseline (Visit 2) of the first drug administration (e.g.; MMR, Varivax).
12. Current alcohol abuse.
13. Current drug abuse or positive drug screen at screening visit. Subjects with legitimate medically supervised uses of the drugs which are not excluded for other reasons (Section 4.2.2 of the protocol) can be enrolled.
14. Patients with any of the following laboratory values at screening and are considered clinically significant by the investigators:

    * Haemoglobin < 9 g/dL, hematocrit, white blood cell count, absolute lymphocyte or platelet count < LLN (below the lower limit of the reference normal range), or absolute neutrophil < 1500/µL
    * ALT, AST and/or total bilirubin > 2 x ULN
    * Serum creatinine > 1.5 x ULN
15. Any clinically significant laboratory abnormalities other than those listed on Exclusion Criteria 14, based on the investigator's medical assessment at screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subject reaching American College of Rheumatology score 20 (ACR20) | at 12-week after the first treatment

SECONDARY OUTCOMES:
Proportion of subjects reaching American College of Rheumatology score 20, 50 and 70 (ACR 20, ACR 50 and ACR70) | up to 24 weeks after the first treatment
Disease Activity Score 28 (DAR28) | up 24 weeks after the first treatment
Target Lesion Psoriasis Severity Score (TLPSS) for subjects with active skin lesions | up 24 weeks after the first treatment
static Physician's Global Assessment (sPGA) for subjects with active skin lesions | up to 24 weeks after the first treatment
Number of subjects with Adverse Event | up to 24 weeks after the first treatment
Immunogenicity | up to 24 weeks after the first treatment
Number of subject with abnormal clinical laboratory parameters | up to 24 weeks after the first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Yao Lin, MD, PhD, Study Director — AbGenomics B.V Taiwan Branch; Mark Genovese, MD, Principal Investigator — Stanford University
Locations (7):
- United States (7):
  - UC San Diego, La Jolla, California
  - Stanford University, Palo Alto, California
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Northwestern University, Chicago, Illinois
  - Justus J. Fiechtner, MD, PC, Lansing, Michigan
  - Metroplex Clinical Research Center, LLC, Dallas, Texas
  - Seattle Rheumatology Associates/Swedish Clinical Research, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No